CLINICAL TRIAL: NCT01596504
Title: An Open-label, Randomized, Three-parallel-group Study on Pharmacodynamic Effects of 8-week QD Treatment With Lixisenatide Compared to Liraglutide in Patients With Type 2 Diabetes Not Adequately Controlled With Insulin Glargine With or Without Metformin
Brief Title: Pharmacodynamic Effects of Lixisenatide Compared to Liraglutide in Patients With Type 2 Diabetes Not Adequately Controlled With Insulin Glargine With or Without Metformin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PDY12625; 2012-000027-40 (EudraCT Number); U1111-1124-1364 (Other: UTN)
Record Dates: First submitted 2012-05-07; First posted 2012-05-11 (Estimated); Results first posted 2016-10-14 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lixisenatide; Liraglutide; Insulin Glargine; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lixisenatide 20 μg (Experimental): Subcutaneous injection of lixisenatide10 μg once daily (QD) for 2 weeks followed by 20 μg QD for 6 weeks under fasted conditions, on top of insulin glargine with or without metformin.
  Interventions: Drug: Lixisenatide (AVE0010); Drug: Insulin Glargine; Drug: Metformin
- Liraglutide 1.2 mg (Active Comparator): Subcutaneous injection of liraglutide 0.6 mg QD for 1 week followed by 1.2 mg QD for 7 weeks under fasted conditions, on top of insulin glargine with or without metformin.
  Interventions: Drug: Liraglutide; Drug: Insulin Glargine; Drug: Metformin
- Liraglutide 1.8 mg (Active Comparator): Subcutaneous injection of liraglutide 0.6 mg QD for 1 week followed by 1.2 mg QD for another 1 week and 1.8 mg QD for next 6 weeks under fasted conditions, on top of insulin glargine with or without metformin.
  Interventions: Drug: Liraglutide; Drug: Insulin Glargine; Drug: Metformin

INTERVENTIONS:
Drug: Lixisenatide (AVE0010) — Pharmaceutical form: solution for injection self-administered with a pen-like injector (OptiClik®).
  Route of administration: subcutaneous
  Arms: Lixisenatide 20 μg
Drug: Liraglutide — Pharmaceutical form:solution for injection
  Route of administration: subcutaneous
  Other Names: Victoza®
  Arms: Liraglutide 1.2 mg; Liraglutide 1.8 mg
Drug: Insulin Glargine — Doses to be adjusted to maintain a fasting self-measured plasma glucose (SMPG) between 4.4 to 5.6 mmol/L (80 to 100 mg/dL)
  Other Names: Lantus® SoloSTAR®
Drug: Metformin — If previously taken metformin to be continued at stable dose throughout the study

SUMMARY:
Primary Objective:

- To investigate the effects of repeated subcutaneous doses of lixisenatide 20 μg once daily (QD) as compared to liraglutide 1.2 mg QD or 1.8 mg QD in reducing post-prandial plasma glucose (PPG) assessed as area under the plasma glucose-concentration-time curve (AUC) after a standardized breakfast at the end of a 8-week treatment period in participants with type 2 diabetes mellitus (T2DM) not adequately controlled with insulin glargine (± metformin).

Secondary Objectives:

* To assess the effects of lixisenatide 20 μg QD as compared to liraglutide 1.2 QD or 1.8 mg QD after an 8-week treatment period in participants with T2DM not adequately controlled with insulin glargine (± metformin) on:

  * Post-prandial C-peptide, glucagon and appetite perceptions after a standardized breakfast,
  * Appetite perceptions after standardized dinner,
  * Gastric emptying after a standardized labelled test meal,
  * Fasting plasma glucose, 24-hour plasma glucose profile,
  * Glycosylated hemoglobin (HbA1c),
  * Insulin glargine dose,
  * 7-point self monitored plasma glucose (SMPG),
  * Body weight and waist circumference,
  * 24-hour heart rate and blood pressure,
* To assess lixisenatide and liraglutide safety and tolerability as add on treatment to insulin glargine (± metformin).

DETAILED DESCRIPTION:
Up to 2-week screening period

* A run-in period of 12 weeks at maximum including a forced titration with insulin glargine up to 11 weeks and 1 baseline pharmacodynamic assessment week
* A 8-week treatment(s) period(s) up to Day 57
* Follow-up: 7 ±2 days after the last treatment day
* Total study duration approximately 14 weeks up to 23 weeks

ELIGIBILITY:
Inclusion criteria :

* Participants with T2DM diagnosed at least 1 year before the screening visit.
* Treatment with neutral protamine hagedorn (NPH) or insulin glargine for at least 3 months and at a stable dose (±20%) of at least 10 IU/day (for at least 2 months prior to screening) alone or combined with a stable dose of metformin with or without dipeptidyl peptidase 4 (DPP-4) inhibitor or sulfonylurea.
* Glycosylated hemoglobin (HbA1c) ≥6.5 and ≤9.5%.
* Body mass index (BMI) between 20 and 40 kg/m^2.

Exclusion criteria:

* Pregnant women or breastfeeding women.
* Clinically relevant history of gastrointestinal disease associated with prolonged nausea and vomiting, including, but not limited to, gastroparesis and gastroesophageal reflux disease requiring medical treatment within 6 months prior to the time of screening.
* Any previous treatment with lixisenatide or participation in a previous study with lixisenatide (AVE0010), and any previous treatment with liraglutide stopped for safety concern or lack of efficacy.
* Allergic reaction to any glucagon-like peptide-1 (GLP-1) agonist in the past (eg, exenatide) or to metacresol.
* History of unexplained pancreatitis, chronic pancreatitis, pancreatectomy, stomach/gastric surgery, inflammatory bowel disease.
* Personal or family history of medullary thyroid cancer (MTC) or a genetic condition that predisposes to MTC.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2012-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (8):
- Germany (8):
  - Investigational Site Number 276008, Berlin
  - Investigational Site Number 276006, Berlin
  - Investigational Site Number 276004, Kiel
  - Investigational Site Number 276002, Mainz
  - Investigational Site Number 276005, Mönchengladbach
  - Investigational Site Number 276007, München
  - Investigational Site Number 276003, Neu-Ulm
  - Investigational Site Number 276001, Neuss

REFERENCES:
- [Result] Meier JJ, Rosenstock J, Hincelin-Mery A, Roy-Duval C, Delfolie A, Coester HV, Menge BA, Forst T, Kapitza C. Contrasting Effects of Lixisenatide and Liraglutide on Postprandial Glycemic Control, Gastric Emptying, and Safety Parameters in Patients With Type 2 Diabetes on Optimized Insulin Glargine With or Without Metformin: A Randomized, Open-Label Trial. Diabetes Care. 2015 Jul;38(7):1263-73. doi: 10.2337/dc14-1984. Epub 2015 Apr 17. PMID 25887358

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 8 centers in Germany between 22 May 2012 to 25 July 2013.
Pre-assignment Details: A total of 236 participants were screened and 142 participants were randomized and treated.
Groups:
- Lixisenatide 20 μg: Subcutaneous injection of lixisenatide10 μg once daily (QD) for 2 weeks followed by 20 μg QD for 6 weeks, on top of insulin glargine with or without metformin.
- Liraglutide 1.2 mg: Subcutaneous injection of liraglutide 0.6 mg QD for 1 week followed by 1.2 mg QD for 7 weeks, on top of insulin glargine with or without metformin.
- Liraglutide 1.8 mg: Subcutaneous injection of liraglutide 0.6 mg QD for 1 week followed by 1.2 mg QD for another 1 week and 1.8 mg QD for next 6 weeks, on top of insulin glargine with or without metformin.
Period: Overall Study
Arm/Group | Lixisenatide 20 μg | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Started | 48 | 47 | 47
Completed | 46 | 44 | 46
Not Completed | 2 | 3 | 1
Not completed — Participant's Private Reason | 0 | 1 | 0
Not completed — Adverse Event | 1 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lixisenatide 20 μg: Subcutaneous injection of lixisenatide10 μg QD for 2 weeks followed by 20 μg QD for 6 weeks, on top of insulin glargine with or without metformin.
- Total: Total of all reporting groups
Arm/Group | Lixisenatide 20 μg | Liraglutide 1.2 mg | Liraglutide 1.8 mg | Total
Number analyzed (Participants) | 48 | 47 | 47 | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (7.4) | 61.4 (7.9) | 62.6 (9.4) | 61.9 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 8 | 14 | 37
  Male | 33 | 39 | 33 | 105
Race [Number; unit: participants]
  Caucasian/White | 48 | 46 | 47 | 141
  Other | 0 | 1 | 0 | 1
Metformin Use at Screening [Number; unit: participants]
  Yes | 43 | 41 | 41 | 125
  No | 5 | 6 | 6 | 17
Weight [Mean (Standard Deviation); unit: kg] | 90.56 (13.09) | 91.62 (13.92) | 92.92 (15.33) | 91.69 (14.07)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: (kg/m²)] | 30.68 (4.34) | 30.52 (4.01) | 31.17 (4.34) | 30.79 (4.22)
HbA1c at Screening (Day -7) [Mean (Standard Deviation); unit: percentage of haemoglobin] | 7.22 (0.48) | 7.19 (0.53) | 7.33 (0.5) | 7.25 (0.50)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 56 in Plasma Glucose Corrected Area Under The Plasma Concentration-Time Curve (AUC) From Time 0.5 Hours to 4.5 Hours
Description: Plasma glucose was assessed using the Gluco-quant Glucose/hexokinase assay. The range of the method was 3 to 1000 milligram per decilitre (mg/dL) with 1 mg/dL as limit of detection (LOD). Calculation of the AUC was made on Day -3 (baseline) and on Day 56 using the linear trapezoidal rule from time of breakfast start (30 minutes after study drug administration [time: 0.5 hours]) to 4 hours after breakfast start (time: 4.5 hours) and corrected by subtracting pre-breakfast plasma glucose concentration (time: 0.5 hours).
Time Frame: 0.5 (prior to standardized breakfast), 0.67, 0.84, 1, 1.5, 2, 2.5, 3.5, 4.5 hours on Day -3 (baseline); 0.5 (prior to standardized breakfast), 0.67, 0.84, 1, 1.5, 2, 2.5, 3.5, 4.5 hours post study drug administration on Day 56
Population: Pharmacodynamic (PD) population defined as all randomized participants, who received at least one dose of lixisenatide 20 μg, liraglutide 1.2 mg or liraglutide 1.8 mg, and had both a baseline assessment and at least one post-baseline assessment of any primary or secondary PD variables, irrespective of compliance with study protocol and procedures.
Measure: Least Squares Mean (Standard Error); unit: h*mmol/L
Arm/Group | Lixisenatide 20 μg | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 43 | 45
h*mmol/L | -13.33 (1.11) | -7.32 (1.12) | -8.72 (1.16)
Statistical Analysis 1: Comparison: Lixisenatide 20 μg vs Liraglutide 1.2 mg; Analysis was performed using linear fixed effects model with treatment groups and stratification factors (HbA1c levels on Day -7 [<8% and >=8%], use of metformin at screening [yes or no]) and the study site) as fixed effects and baseline plasma glucose AUC from 0.5 to 4.5 hours as covariate. To address multiplicity issue and ensure overall 1-sided level of 5%, Hochberg method was used for testing procedure of comparison between lixisenatide vs liraglutide 1.2 mg or 1.8 mg; Test type: Superiority or Other; p < 0.0001, Linear fixed effects model — p-values ordered(p1≤p2) as per rules:if p2≤0.05: lixisenatide superior to liraglutide (both doses);if p2>0.05 & p1≤0.025:lixisenatide superior to dose of liraglutide associated with p1;if p2>0.05 & p1>0.025:no comparison as statistically significant; The threshold for significance at 0.05 level; Least squares (LS) mean difference = -6.01, 95% CI 1-sided [lower limit -7.77], Standard Error of Mean 1.06 — Lixisenatide vs Liraglutide 1.2 mg
Statistical Analysis 2: Comparison: Lixisenatide 20 μg vs Liraglutide 1.8 mg; Analysis was performed using linear mixed effects model with treatment groups and stratification factors (HbA1c levels on Day -7 [<8% and >=8%], use of metformin at screening [yes or no]), and the study site) as fixed effects and baseline plasma glucose AUC from 0.5 to 4.5 hours as covariate. To address multiplicity issue and ensure overall 1-sided level of 5%, Hochberg method was used for testing procedure of comparison between lixisenatide vs liraglutide 1.2 mg or 1.8 mg; Test type: Superiority or Other; p < 0.0001, Linear fixed effects model — p-values ordered(p1≤p2) as per rules:if p2≤0.05:lixisenatide superior to liraglutide (both doses);if p2>0.05 & p1≤0.025:lixisenatide superior to dose of liraglutide associated with p1;if p2>0.05 & p1>0.025: no comparison as statistically significant; The threshold for significance at 0.05 level; LS mean difference = -4.61, 95% CI 1-sided [lower limit -6.34], Standard Error of Mean 1.04 — Lixisenatide vs Liraglutide 1. 8 mg

2. Secondary Outcome: Change From Baseline to Day 56 in Plasma Glucose Corrected AUC From Time 0.5 Hours to 5.5 Hours
Description: Plasma glucose was assessed using the Gluco-quant Glucose/hexokinase assay. The range of the method was 3 to 1000 mg/dL with 1 mg/dL as limit of detection (LOD). Calculation of the AUC was made on Day -3 (baseline) and on Day 56 using the linear trapezoidal rule from time of breakfast start (30 minutes after study drug administration [time: 0.5 hours]) to 5 hours after breakfast start (time: 5.5 hours) and corrected by subtracting pre-breakfast plasma glucose concentration (time: 0.5 hours).
Time Frame: 0.5 (prior to standardized breakfast), 0.67, 0.84, 1, 1.5, 2, 2.5, 3.5, 4.5, 5.5 hours on Day -3 (baseline); 0.5 (prior to standardized breakfast), 0.67, 0.84, 1, 1.5, 2, 2.5, 3.5, 4.5, 5.5 hours post study drug administration on Day 56
Population: PD population. Number of participants analyzed = participants with plasma glucose assessment at specified time-points.
Measure: Least Squares Mean (Standard Error); unit: h*mmol/L
Groups:
- Lixisenatide 20 µg: Subcutaneous injection of lixisenatide10 μg QD for 2 weeks followed by 20 μg QD for 6 weeks, on top of insulin glargine with or without metformin.
Arm/Group | Lixisenatide 20 µg | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 43 | 45
h*mmol/L | -13.82 (1.19) | -9.09 (1.21) | -10.33 (1.25)

3. Secondary Outcome: Number of Participants With 2-Hour Post-prandial Plasma Glucose (PPG) <7.77 (mmol/L) at Day 56
Description: Plasma glucose was assessed using the Gluco-quant Glucose/hexokinase assay. The range of the method was 3 to 1000 mg/dL with 1 mg/dL as LOD. The 2-hour PPG test measured blood glucose 2 hours after start of a standardised breakfast.
Time Frame: Day 56
Population: PD population. Number of participants analyzed = participants with plasma glucose assessment at specified time-points.
Measure: Number; unit: participants
Arm/Group | Lixisenatide 20 µg | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 44 | 46
participants | 35 | 13 | 11

4. Secondary Outcome: Change From Baseline to Day 56 in PPG Excursion
Description: Plasma glucose was assessed using the Gluco-quant Glucose/hexokinase assay. The range of the method was 3 to 1000 mg/dL with 1 mg/dL as LOD. PPG excursion was determined on Day -3 (Baseline) and Day 56 as the maximum change in PPG from time of breakfast start (time: 0.5 hours) until 5 hours later (time: 5.5 hours) subtracted from pre-meal plasma concentration.
Time Frame: 0.67, 0.84, 1, 1.5, 2, 2.5, 3.5, 4.5, 5.5 hours on Day -3 (baseline); 0.67, 0.84, 1, 1.5, 2, 2.5, 3.5, 4.5, 5.5 hours post study drug administration on Day 56
Population: PD population. Number of participants analyzed = participants with plasma glucose assessment at specified time-points.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lixisenatide 20 µg | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 43 | 45
mmol/L | -3.26 (0.4) | -1.79 (0.4) | -2.5 (0.42)

5. Secondary Outcome: Change From Baseline to Day 56 in Fasting Plasma Glucose (FPG)
Description: Plasma glucose was assessed using the Gluco-quant Glucose/hexokinase assay. The range of the method was 3 to 1000 mg/dL with 1 mg/dL as LOD. The value of FPG on Day -3 was the baseline.
Time Frame: 0.5 hour (prior to standardized breakfast) on Day -3; 0.5 hour (prior to standardized breakfast) on Day 56
Population: PD population. Number of participants analyzed = participants with plasma glucose assessment at specified time-points.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lixisenatide 20 µg | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 45 | 44 | 45
mmol/L | 0.1 (0.22) | 0.12 (0.22) | 0.13 (0.23)

6. Secondary Outcome: Change From Baseline to Day 56 in Average 7-Point Self-Monitored Plasma Glucose (SMPG)
Description: Seven-point SMPG (before breakfast, 2 hours post breakfast, before lunch, 2 hours post lunch, before dinner, 2 hours post dinner, and at bedtime) was measured using Freestyle Precision glucometer and average of the 7 measurements was calculated.
Time Frame: Before breakfast, 2 hours post breakfast, before lunch, 2 hours post lunch, before dinner, 2 hours post dinner, and at bedtime on Day -3 (Baseline) and on Day 56
Population: PD population. Number of participants analyzed = participants with 7 point SMPG assessment at specified time-points.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lixisenatide 20 µg | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 44 | 46
mmol/L | -0.69 (1.19) | -0.76 (1.23) | -1.2 (1.09)

7. Secondary Outcome: Change From Baseline to Day 56 in Corrected C-Peptide AUC From Time 0.5 Hours to 5.5 Hours
Description: C-peptide was assessed using the Electro Chemiluminescence Immuno Assay.The range of the method was 0.2 to 25 nanogram per millilitre (ng/mL) and the LOD was 0.07 ng/mL. Measurement was done on Day -3 (Baseline) and Day 56 as the maximum change in C-peptide from time of breakfast start (time: 0.5 hours) until 5 hours later (time: 5.5 hours) subtracted from pre-meal plasma concentration.
Time Frame: 0.5 (prior to standardized breakfast), 0.67, 0.84, 1, 1.5, 2, 2.5, 3.5, 4.5, 5.5 hours on Day-3 (baseline); 0.5 (prior to standardized breakfast), 0.67, 0.84, 1, 1.5, 2, 2.5, 3.5, 4.5, 5.5 hours post study drug administration on Day 56
Population: PD population. Number of participants analyzed = participants with C-peptide assessment at specified time-points.
Measure: Least Squares Mean (Standard Error); unit: h*nmol/L
Arm/Group | Lixisenatide 20 µg | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 43 | 45
h*nmol/L | -1.16 (0.37) | 1.23 (0.37) | 0.88 (0.39)

8. Secondary Outcome: Change From Baseline to Day 56 in Corrected Glucagon AUC From Time 0.5 Hours to 5.5 Hours
Description: Glucagon was assessed using the radioimmunoassay. The range of the method was 4.7 to 150 picomole per litre (pmol/L). Measurement was done on Day -3 (Baseline) and Day 56 as the maximum change in glucagon from time of breakfast start (time: 0.5 hours) until 5 hours later (time: 5.5 hours) subtracted from pre-meal plasma concentration.
Time Frame: 0.5 (prior to standardized breakfast), 0.67, 0.84, 1, 1.5, 2, 2.5, 3.5, 4.5, 5.5 hours on Day -3 (baseline); 0.5 (prior to standardized breakfast), 0.67, 0.84, 1, 1.5, 2, 2.5, 3.5, 4.5, 5.5 hours post study drug administration on Day 56
Population: PD population. Number of participants analyzed = participants with glucagon assessment at specified time-points.
Measure: Least Squares Mean (Standard Error); unit: h*ng/L
Arm/Group | Lixisenatide 20 µg | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 43 | 45
h*ng/L | -16.56 (19.43) | 11.58 (19.86) | 5.6 (20.3)

9. Secondary Outcome: Change From Baseline to Day 56 in HbA1c
Description: HbA1C was assessed using the high performance liquid chromatography method.
Time Frame: Pre-dose (Hour 0) on Day 1 (Baseline) and Day 56
Population: Number of participants analyzed = participants with HbA1c assessment at specified time-points.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Lixisenatide 20 µg | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 44 | 46
percentage of HbA1c | -0.58 (0.06) | -0.66 (0.06) | -0.74 (0.06)

10. Secondary Outcome: Change From Baseline to Day 56 in Average Daily Insulin Glargine Dose
Time Frame: Day -7 (Baseline), Day 56
Population: PD population. Number of participants analyzed=participants with insulin glargine dose assessment at specified time-points.
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Lixisenatide 20 µg | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 44 | 46
units | -4.7 (4.8) | -4.6 (6.8) | -4.0 (6.5)

11. Secondary Outcome: Change From Baseline to Day 55 in Gastric Emptying Half Life (t1/2)
Description: Gastric emptying was measured using 13C-octanoic acid breath test by isotope-selective non-dispersive infrared spectrometry.
Time Frame: 0 (prior to standardized breakfast), 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5, 4, 4.5, 5, 5.5 hours on Day -4 (baseline) and on Day 55
Population: PD population. Number of participants analyzed=participants with gastric emptying assessment at specified time-points.
Measure: Least Squares Mean (Standard Error); unit: minutes (min)
Arm/Group | Lixisenatide 20 µg | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 44 | 46
minutes (min) | 453.56 (58.24) | 175.31 (58.49) | 130.49 (60.27)

12. Secondary Outcome: Change From Baseline to Day 55 in Gastric Emptying Coefficient
Description: Gastric emptying was measured using 13C-octanoic acid breath test by isotope-selective non-dispersive infrared spectrometry. Gastric emptying coefficient was derived from a mathematical formula that describes the gastric emptying rate and gives an overall index of gastric emptying.
Time Frame: 0 (7:30 clock time, prior to standardized breakfast), 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3, 3.5, 4, 4.5, 5, 5.5 hours on Day -4 (baseline) and on Day 55
Population: PD population. Number of participants analyzed = participants with gastric emptying at specified time-points.
Measure: Mean (Standard Deviation); unit: coefficient (unit-less)
Arm/Group | Lixisenatide 20 µg | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 44 | 46
coefficient (unit-less) | -0.33 (1.09) | -0.34 (0.53) | -0.28 (0.52)

13. Secondary Outcome: Change From Baseline to Day 57/58 in 24-Hour Mean Heart Rate
Description: The baseline value was the 24-hour mean on Day -2/-1 determined as overall, night and daytime mean. Measurements were made every 15 minutes from 07:00 to 23:00 (daytime) and every 30 minutes from 23:00 to 07:00 (night-time) at baseline and Day 57/58. Measurements were obtained after 10 minutes in the supine resting position.
Time Frame: Every 15 minutes from 07:00 clock time to 23:00 clock time (day-time) and every 30 minutes from 23:00 clock time to 07:00 clock time (night-time) on Day -2/-1 (Baseline) and Day 57/58
Population: PD population. Number of participants analyzed = participants with heart rate assessment at specified time-points.
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | Lixisenatide 20 µg | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 42 | 43 | 44
beats per minute | 3.34 (1.33) | 9.33 (1.24) | 9.17 (1.31)

14. Secondary Outcome: Change From Baseline to Day 57/58 in 24-Hour Mean Systolic Blood Pressure and Diastolic Blood Pressure
Description: The baseline value was the 24-hour means on Day -2/-1 determined as overall, night and day-time mean. Measurements were made every 15 minutes from 07:00 to 23:00 (day-time) and every 30 minutes from 23:00 to 07:00 (night-time) at baseline and at Day 57/58. Measurements were obtained after 10 minutes in the supine resting position.
Time Frame: Every 15 minutes from 07:00 clock time to 23:00 clock time (day-time) and every 30 minutes from 23:00 clock time to 07:00 clock time (night-time) on Day -2/ -1 (Baseline) and Day 57/58
Population: PD population. Number of participants analyzed = participants with blood pressure assessment at specified time-points.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lixisenatide 20 µg | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 42 | 43 | 44
mmHg
  24-Hour Mean Systolic Blood Pressure | 0.4 (6.4) | -0.5 (7.1) | -2.5 (7.7)
  24-Hour Mean Diastolic Blood Pressure | 0.8 (4.1) | 2.4 (4.7) | 1.6 (4.7)

15. Secondary Outcome: Change From Baseline to Day 57 in Body Weight
Time Frame: 0.5 hours prior to standardized breakfast on Day -1 (Baseline); 0.5 hours prior to study drug administration on Day 57
Population: PD population. Number of participants analyzed = participants with body weight assessment at specified time-points.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Lixisenatide 20 µg | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 44 | 46
kg | -1.61 (0.47) | -1.78 (0.48) | -2.42 (0.49)

16. Secondary Outcome: Change From Baseline to Day 57 in Waist Circumference
Time Frame: 0.5 hours prior to standardized breakfast on Day -1 (Baseline); 0.5 hours prior to IMP administration on Day 57
Population: PD population. Number of participants analyzed = participants with waist circumference assessment at specified time-points.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Lixisenatide 20 µg | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 43 | 46
cm | -1.40 (4.66) | -1.93 (3.59) | -2.12 (4.95)

17. Secondary Outcome: Change From Baseline to Day 56 in the Cumulative Score Mean on the Appetite Perception Using a Visual Analogue Scale After Standardized Solid Breakfast
Description: Visual Analogue Scale, 100 mm in length with words anchored at each end, expressing the most positive (100 mm) and the most negative rating (0 mm), was used to assess hunger, satiety, fullness and prospective food consumption. Responses were measured as distance from the left end of the line to the mark. Mean change from baseline was calculated for each parameter separately.
Time Frame: 0.5 (8:00 clock time, prior to standardized breakfast), 1.5, 2.5, 3.5, 4.5, 5.5 hours on Day -3; 0 (prior to standardized breakfast), 1.5, 2.5, 3.5, 4.5, 5.5 hours post study drug administration on Day 56
Population: PD population. Number of participants analyzed=participants with appetite perception assessment at specified time-points.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Lixisenatide 20 µg | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 44 | 46
mm
  How hungry do you feel? | -3.7 (16.4) | -3.1 (16.8) | -1.0 (14.6)
  How satisfied do you feel? | 4.5 (15.8) | 8.9 (13.2) | 3.6 (11.0)
  How full do you feel? | 4.9 (17.0) | 9.3 (15.6) | 6.4 (13.8)
  How much do you think you can eat? | -6.4 (16.1) | -4.5 (15.7) | -7.2 (12.0)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the end of study (10 weeks) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent adverse events that developed/worsened during the 'on treatment period' (the time from the first drug injection [included] up to 3 days after the last injection of drug administration [included]).
Arm/Group | Lixisenatide 20 µg | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Serious Adverse Events (participants affected / at risk) | 1/48 | 1/47 | 0/47
Other Adverse Events (participants affected / at risk) | 26/48 | 27/47 | 27/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lixisenatide 20 µg (N=48) | Liraglutide 1.2 mg (N=47) | Liraglutide 1.8 mg (N=47)
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lixisenatide 20 µg (N=48) | Liraglutide 1.2 mg (N=47) | Liraglutide 1.8 mg (N=47)
Abdominal distension (Gastrointestinal disorders) | 3 | 7 | 4
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 5
Constipation (Gastrointestinal disorders) | 0 | 5 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 5
Dyspepsia (Gastrointestinal disorders) | 3 | 3 | 4
Flatulence (Gastrointestinal disorders) | 2 | 0 | 4
Nausea (Gastrointestinal disorders) | 9 | 8 | 11
Vomiting (Gastrointestinal disorders) | 5 | 2 | 5
Fatigue (General disorders) | 3 | 1 | 4
Malaise (General disorders) | 3 | 0 | 1
Nasopharyngitis (Infections and infestations) | 6 | 10 | 5
Decreased appetite (Metabolism and nutrition disorders) | 9 | 9 | 13
Dizziness postural (Nervous system disorders) | 3 | 1 | 0
Headache (Nervous system disorders) | 4 | 5 | 8
Insomnia (Psychiatric disorders) | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months after trial completion, the Investigator can present or publish results. The investigator provides the sponsor with a copy of the presentation or publication for review and comment at least 30 days in advance of its submission.

The sponsor can delay the submission for a period not exceeding 90 days to allow for filing a patent application or such other measures as sponsor deems appropriate to establish and preserve its proprietary rights.